CLINICAL TRIAL: NCT03363230
Title: Effects of Mindfulness Training on Emotion Regulation and Impulsivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Principal Investigator, Juan Carlos Pascual, Principal Investigator, Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIBSP-TLP-2013-115
Record Dates: First submitted 2017-11-30; First posted 2017-12-06 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-11

CONDITIONS: Mindfulness Skills; Interpersonal Effectiveness Skills
Keywords: mindfulness; emotion regulation; impulsivity
MeSH Terms: conditions — Emotional Regulation; Impulsive Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness skills (Experimental)
  Interventions: Behavioral: Mindfulness skills training
- Interpersonal effectiveness skills (Active Comparator)
  Interventions: Behavioral: Interpersonal Effectiveness skills training

INTERVENTIONS:
Behavioral: Mindfulness skills training — Mindfulness skills were taught over a 10-week period. Mindfulness skills were delivered in a weekly group-format. Participants were instructed to follow mindfulness practice at home. The treatment was focused on enhancing the patient capacity to defuse from cognitive and emotional content.
  Arms: Mindfulness skills
Behavioral: Interpersonal Effectiveness skills training — Interpersonal effectiveness skills were taught over a 10-week period. Skills were delivered in a weekly group-format. The treatment was focused on improving interpersonal effectiveness.
  Arms: Interpersonal effectiveness skills

SUMMARY:
Mindfulness training has proven to be a reliable treatment for patients with Borderline Personality Disorder (BPD).The present randomized-controlled study examines the effects of mindfulness training on emotion regulation and impulsitivy. In addition, fMRI data was collected pre and post intervention. 70 patients with BPD diagnosis were randomized to either mindfulness or interpersonal effectiveness skills training. Assessments were conucted pre-and-post-intervention.

ELIGIBILITY:
Inclusion criteria:

* BPD diagnosis according to two semi -structured interviews: the Structured Clinical Interview for DSM-IV Axis II disorders and the Revised Diagnostic Interview for Borderlines
* Age between 18 and 50 years old
* No comorbidities with schizophrenia, drug induced psychosis, organic brain syndrome, substance dependence, bipolar disorder, mental retardation, or major depressive episode in course
* Not being participating in any other psychotherapy at the moment of the study.

Exclusion criteria:

• Having participated of skills training in the past.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Difficulties in Emotion Regulation Scale (DERS) | 1-past week
  The DERS is a 28-item-scale that measures difficulties in emotion regulation. Each item has to be rated in a 5-point scale, with higher scores indicating higher difficulties in emotion regulation.
Barrat Impulsiveness Scale (BIS-11) | 1-past week
  The current version of the Barratt Impulsiveness Scale is composed of 30 items describing common impulsive or non-impulsive (for reverse scored items) behaviors and preferences. Items are scored on a 4-point-scale, with higher scores indicating higher impulsivity.

SECONDARY OUTCOMES:
Borderline Symptoms List (BSL-23) | 1-past-week
  The BSL-23 assess common borderline symptoms during the past week (higher scores indicating higher borderline features). Items have to be rated on a 5-point-scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Storebo OJ, Stoffers-Winterling JM, Vollm BA, Kongerslev MT, Mattivi JT, Jorgensen MS, Faltinsen E, Todorovac A, Sales CP, Callesen HE, Lieb K, Simonsen E. Psychological therapies for people with borderline personality disorder. Cochrane Database Syst Rev. 2020 May 4;5(5):CD012955. doi: 10.1002/14651858.CD012955.pub2. PMID 32368793